CLINICAL TRIAL: NCT00258505
Title: Incidence, Nature and Consequences of Cortical Depolarizations in Human Brain Injury From Trauma and Ischemia: The COSBID Study
Brief Title: Monitoring Brain Activity in Human Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Other Study IDs: sor402605ctil
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2005-10

CONDITIONS: Traumatic Brain Injury; Aneurysmal Subarachnoid Hemorrhage; Cerebral Infarction; Cerebral Hemorrhage
Keywords: Spreading depression; Seizures; Blood-brain barrier
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Cerebral Infarction; Cerebral Hemorrhage; Seizures

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Procedure: intracranial monitoring up to 9 days after injury

SUMMARY:
The outcome of brain injury (physical or stroke) may be related to a brain electrical phenomenon known as Cortical Spreading Depression (CSD). This is a brief cessation of function in a local region of brain tissue. It has been hypothesized that CSD may occur after brain injury and may expand the damage to adjacent brain areas. Our aim is to detect CSD by means of intracranial electrodes in patients with brain injuries and asses how these events alter the outcome of the patients.

DETAILED DESCRIPTION:
Cortical spreading depression (CSD) is a wave of mass neuronal firing and neuronal and glial depolarisation which propagates through grey matter in the central nervous system in response to a pathologic stimulus, at a rate of between 1 and 5 mm per minute. First described by Leão in 1944 as a sudden depression of ECoG amplitude spreading across the cortex of the rabbit (Leao, A. A. P. 1944), CSD can be elicited in experimental animals by chemical, electrical, and mechanical stimuli, with varying degrees of ease. CSD provoked in healthy, normally perfused neural tissue does not induce persistent metabolic stress or cellular damage, and indeed such induction of CSD in animal experiments may confer protection against the adverse effects of a subsequent ischaemic insult (Kobayashi, S. et al. 1995).

In animal models of focal cerebral ischaemia, usually induced by occlusion of the middle cerebral artery, a spontaneous phenomenon occurs around the periphery of the core territory, with electrophysiological features essentially identical with CSD, and similar capacity to propagate across cerebral cortex. Designated "peri-infarct depolarisation" (PID), this event is associated with infarct expansion, or recruitment of at-risk cortical territory into the expanding core, and has been shown capable of causing this expansion, in the absence of therapeutic intervention. Indeed it has been hypothesized that glutamate release may be involved in PID generation, and that excitotoxicity may accomplish detrimental effects via this route (Hossmann, K. A. 1994), (Obrenovitch, T. P. and Urenjak, J. 1997). Some experimental neuroprotection treatments for stroke act to decrease the incidence of PID (Iijima, T. et al. 1992;Chen, Q. et al. 1993;Busch, E. et al. 1996).

In traumatic and ischaemic (especially in middle cerebral artery occlusion and aneurysmal subarachnoid haemorrhage) brain injury in humans, a phase of delayed deterioration often associated with severe and refractory brain swelling develops between 2 and 5 days after the initial ictus, and is associated with poor or fatal outcome. The cause and mechanism of this deterioration remain poorly understood, and the possibility exists that CSD/PID events might contribute to deterioration.

To date, CSD or PID have been reported in only ten human subjects in two papers (Mayevsky, A. et al. 1996; Strong, A. J. et al. 2002). Strong et al. reported that transient ECoG suppressions suggestive of depolarisations are common - but by no means universal - after brain injury in humans. Sub-dural ECoG electrode strips were placed in 14 patients who had undergone craniotomy for trauma or intracranial hemorrhage; monitoring was for up to 60 h following the injury. Five of these patients (36%) showed patterns of ECoG depression consistent with PID/CSD in brain regions adjacent to the primary injury.

ELIGIBILITY:
Inclusion Criteria:

Immediately following:

* traumatic brain injury
* aneurysmal subarachnoid haemorrhage or
* spontaneous intracerebral haematoma or
* stroke involving cerebral cortex

Exclusion Criteria:

* GCS = 3
* Bilateral fixed & dilated pupils or other evidence of massive irreversible brain injury
* more than 5 days post Injury/ictus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Study Completion 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Alon Friedman, MD/PhD, Principal Investigator — Soroka University Medical Center; Jens Dreier, MD, Principal Investigator — Charite, Berlin, Germany
Locations (2):
- Charite, Berlin, Germany
- Soroka, Beersheba, Israel

REFERENCES:
- [Background] Strong AJ, Fabricius M, Boutelle MG, Hibbins SJ, Hopwood SE, Jones R, Parkin MC, Lauritzen M. Spreading and synchronous depressions of cortical activity in acutely injured human brain. Stroke. 2002 Dec;33(12):2738-43. doi: 10.1161/01.str.0000043073.69602.09. PMID 12468763
- See also: For List of Participants see http://www.cosbid.org/ — http://www.cosbid.org/